CLINICAL TRIAL: NCT01584531
Title: A Phase II, Multicenter, Single-arm Study to Assess the Efficacy and Safety of Oral Rigosertib in Transfusion-dependent Low or Intermediate-1 (Any Cytogenetics) or Trisomy 8 Intermediate-2 Myelodysplastic Syndrome Patients Based on IPSS Classification
Brief Title: Efficacy and Safety of Oral Rigosertib in Transfusion-dependent, Low or Int-1 or Trisomy 8 Int-2 Myelodysplastic Syndrome
Acronym: ONTARGET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 09-05; AAAJ0151 (Other: Columbia University)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Myelodysplastic Syndrome; MDS; Trisomy 8
Keywords: rigosertib sodium; rigosertib; ON 01910.Na; oral rigosertib
MeSH Terms: conditions — Myelodysplastic Syndromes; Chromosome 8, trisomy | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 21-Day Regimen (Experimental): 560 mg oral rigosertib in the morning and 280 mg rigosertib in the afternoon on days 1 to 21 of 21-day cycle
  Interventions: Drug: rigosertib

INTERVENTIONS:
Drug: rigosertib — Rigosertib sodium will be available as soft gel capsules in strengths of 280 mg and 70 mg. Rigosertib will be administered on an outpatient basis.
  Patients will take a 560 mg dose (e.g., 2 x 280 mg capsules) of oral rigosertib in the morning and 280 mg dose (e.g., 1 x 280 mg capsules) of oral rigosertib every day of 21-day cycles. Rigosertib should be taken in a fasting state (defined by at least 30 minutes before next meal) BID at 12 hr intervals (with a window of 2 hr). Any vomited dose will be reported as a missed dose.
  The patient will fill a diary indicating the day and time of drug intake.
  Other Names: rigosertib sodium; ON 01910.Na; oral rigosertib

SUMMARY:
The primary objectives of this study are to determine if rigosertib sodium, given orally in the form of soft gel capsules, is safe and is associated with a reduction in the number of blood transfusion units that are needed in patients with myelodysplastic syndrome (MDS) classified as Low or Intermediate-1 (Int-1) (any cytogenetics) or trisomy 8 Intermediate 2 (Int-2) in the International Prognostic Scoring System (IPSS) who are transfusion-dependent. Rigosertib will be taken on days 1 to 21 of a 21-day cycle.

DETAILED DESCRIPTION:
This will be a Phase II open-label, multicenter (up to 5 centers), single-arm study. Sixty transfusion-dependent patients with MDS classified as Low or Int-1 risk (any cytogenetics) or trisomy 8 Int-2 by International Prognostic Scoring System (IPSS) will be enrolled to receive rigosertib BID for 21 consecutive days of a 21-day cycle.

Patients will be stratified on prior treatment with azacitidine and/or decitabine and/or lenalidomide and/or erythropoietin.

Patients will remain treated on study until 2006 Internation Working Group (IWG) progression criteria are met or until death from any cause.

All study participants will be allowed, as medically justified, access to RBC and platelet transfusions, and to filgrastim [G-CSF]. Erythropoiesis-stimulating agents (ESAs) will not be allowed during the initial 3 cycles. Rigosertib dosing adjustment policies are described in Protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS confirmed by bone marrow aspirate and/or biopsy within 6 weeks prior to first dose of study drug according to World Health Organization (WHO) or French-American-British (FAB) classification
* MDS classified as Low risk or Int-1 risk (any cytogenetics) or Trisomy 8 Int-2 risk, according to IPSS classification
* Transfusion dependency defined by at least 4 units of RBC administered within 8 weeks before baseline
* Off all other treatments for MDS (azacitidine, decitabine, lenalidomide, chemotherapy, immunosuppressive agents) for at least 4 weeks
* ECOG performance status of 0, 1 or 2

Exclusion Criteria:

* Ongoing clinically significant anemia due to factors such as iron, B12, or folate deficiencies, auto-immune or hereditary hemolysis, or gastrointestinal (GI) bleeding, unless stabilized for 1 week after RBC transfusion
* Serum ferritin <50 ng/mL
* Hypoplastic MDS (cellularity <10%)
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Active infection not adequately responding to appropriate therapy
* Total bilirubin ≥1.5 mg/dL not related to hemolysis or Gilbert's disease
* ALT/AST ≥2.5 x upper limit of normal (ULN)
* Serum creatinine ≥2.0 mg/dL
* Ascites requiring active medical management including paracentesis
* Hyponatremia (defined as serum sodium value of <130 mEq/L)
* Female patients who are pregnant or lactating
* Patients who are unwilling to follow strict contraception requirements
* Female patients with reproductive potential who do not have a negative urine beta-human chorionic gonadotropin (bHCG) pregnancy test at Screening
* Major surgery without full recovery or major surgery within 3 weeks of rigosertib treatment start
* Uncontrolled hypertension (defined as a systolic pressure ≥160 mmHg and/or a diastolic pressure ≥110 mmHg)
* New onset seizures (within 3 months prior to the first dose of rigosertib) or poorly controlled seizures
* Any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy
* Chronic use (>2 weeks) of corticosteroids (>10 mg/24 hr equivalent prednisone) within 4 weeks of starting rigosertib
* Investigational therapy within 4 weeks of starting rigosertib
* Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of units of red blood cell transfusions | 8 weeks
  Number of units of red blood cell transfusions will be compared with the pretreatment transfusion number in the previous 8 weeks.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | From date of randomization until 30 days after last dose of study drug
  AEs reported by the patient or observed by the Investigator or study site personnel Safety assessments will be counted and documented on Case Report Forms and source documents. All AEs from signature of the ICF through 30 days after a patient discontinues from the study will be included.
Bone marrow blasts | 4 weeks
  Change in number of bone marrow blasts will be compared to pretreatment.
Complete blood count | 4 weeks
  Complete blood count with differential.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Fruchtman, MD, Study Director — Traws Pharma, Inc.
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Bon Secours St. Francis Hospital, Greenville, South Carolina

REFERENCES:
- [Background] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: The Leukemia & Lymphoma Society — http://www.lls.org/
- See also: The Myelodysplastic Syndromes Foundation — http://www.mds-foundation.org/